CLINICAL TRIAL: NCT05431088
Title: A Phase 2/3 Randomized, Multicenter Study of Osivelotor Administered Orally to Adult and Adolescent Participants With Sickle Cell Disease
Brief Title: A Phase 2/3 Study in Adult and Adolescent Participants With SCD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GBT021601-021; C5351004 (Other: Alias Study Number); 2023-508766-14-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part B only
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A (Active Comparator): Initially, participants will be randomized 1:1 to 100 mg and 150 mg daily. Upon review of the 150 mg safety data from at least 6 participants, there will be 1:1:1 randomization: 100 mg, 150 mg, and up to 200 mg.
  Participants will then receive maintenance once daily doses through Week 12.
  Interventions: Drug: Osivelotor
- Part B (Placebo Comparator): Study drug arm: Adult participants will receive osivelotor at 300 mg QD loading dose for 7 days followed by 150 mg QD through Week 48.
  Adolescent participant dose will be defined in a future protocol amendment.
  Placebo arm: Participants will receive placebo tablets for 48 weeks.
  Interventions: Drug: Osivelotor
- OLE (Experimental): Adult Participants will receive 150 mg open-label osivelotor up to 2 years after the last participant's visit in Part B or when the drug is commercially available in that region.
  The appropriate doses for adolescents will be defined in a future protocol amendment.
  Interventions: Drug: Osivelotor

INTERVENTIONS:
Drug: Osivelotor — Tablets which contain drug substance
  Other Names: PF-07940367 or GBT021601

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of osivelotor.

DETAILED DESCRIPTION:
This is a three-part, multicenter, Phase 2/3 study of orally administered osivelotor in participants with sickle cell disease (SCD).

Part A will evaluate the safety, tolerability, and efficacy of osivelotor in adult participants with SCD to determine an optimal dose.

Part B will evaluate the efficacy of osivelotor versus placebo in adult and adolescent participants with SCD for 48 weeks.

Open Label Extension (OLE) will evaluate the long-term safety and hematologic responses of open-label osivelotor in adult and adolescent participants having completed Part B.

ELIGIBILITY:
Inclusion Criteria:

Part A, Part B, and OLE:

* Male or female with SCD
* Participants with stable Hb value as judged by the Investigator
* For participants taking hydroxyurea and/or L-glutamine, the dose must be stable for at least 90 days prior to signing the ICF or assent and with no anticipated need for dose adjustments during the study in the opinion of the Investigator.

Part B:

* Participants with SCD ages 12 to 65 years, inclusive
* Participants with more than or equal to 2 and ≤ 10 VOCs within 12 months of Screening.

OLE:

- Participants who have completed the Part B will be eligible.

Exclusion Criteria:

Part A, Part B, and OLE:

* Participants who had more than 10 VOC within 12 months of screening
* Female participant who is breastfeeding or pregnant
* Participants who receive RBC transfusion therapy regularly or received an RBC transfusion ---for any reason within 90 days of Day 1
* Participants hospitalized for sickle cell crisis or other vaso-occlusive event within 14 days of signing the ICF or anytime during the screening period.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 389 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A | Through week 12
  Number of adult participants with change from baseline in hemoglobin (Hb) through week 12 as measured by change in osivelotor concentrations from baseline or percentage change from baseline of clinical measures of anemia Hb and hemolysis (including indirect bilirubin, reticulocytes and lactate dehydrogenase).
Part B | Through week 48
  Co-primary endpoints: Hb response (increase from baseline of >1 g/dL) at Week 48 (based on average of Hb levels at Week 40 and Week 48) and the Annualized rate of VOC through end of Week 48.
  A VOC is defined as an acute episode of pain that:
  * Has no medically determined cause other than a vaso-occlusive event, and
  * Results in a visit to a medical facility (hospitalization, emergency department, urgent care center, outpatient clinic, or infusion center), and
  * Requires parenteral narcotic agents, parenteral nonsteroidal anti-inflammatory drugs (NSAIDs), or an increase in treatment with oral narcotics.
  Complicated VOCs of acute chest syndrome (ACS), hepatic sequestration, splenic sequestration, priapism, and dactylitis that meet the requirements listed above will be included in this co-primary endpoint.
OLE | Approximately 24 months after last patient enrolled
  Incidence of Treatment Emergent Adverse Events:
  * Incidence of SAEs
  * Incidence of AEs leading to discontinuation
  * Change from baseline in laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (22):
  - Smilow Cancer Hospital, New Haven, Connecticut
  - Children's National Hospital, Washington D.C., District of Columbia
  - Edward Jenner Research Group Center LLC, Plantation, Florida
  - Pediatric Hematology / Oncology a division of Kidz Medical services, West Palm Beach, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Alpha Clinical Research Georgia, Dunwoody, Georgia
  - Sonar Clinical Research, Riverdale, Georgia
  - University of Illinois at Chicago Clinical Research Center, Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System - Investigational Drug Services (IDS), Chicago, Illinois
  - University of Illinois Hospital and Health Sciences System, Chicago, Illinois
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Hospital, Inc., Baton Rouge, Louisiana
  - Our lady of the Lake Hospital, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - University Health, Kansas City, Missouri
  - UNC Health, Chapel Hill, North Carolina
  - McGovern Medical School at UTHealth, Houston, Texas
  - Memorial Hermann Hospital, Texas Medical Center - Clinical Research Unit (CRU), Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - UT Physicians Comprehensive Sickle Cell Clinic, Houston, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Brazil (9):
  - Hospital Universitario Professor Edgar Santos, Salvador, Estado de Bahia
  - Multihemo Servicos Medicos S/A, Recife, Pernambuco
  - Hospital Das Clinicas da Faculdade de Medicina de Ribeirão Preto - USP, Ribeirão Preto, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Casa de Saude Santa Marcelina, São Paulo, São Paulo
  - Instituto Estadual de Hematologia Arthur Siqueira Cavalcanti - HEMORIO, Rio de Janeiro
  - Esho Empresa De Servicos Hospitalares S.A/ Hospital Samaritano Higienopolis, São Paulo
  - Real e Benemerita Associacao Portuguesa de Sao Paulo, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
- India (2):
  - Nirmal Hospital Pvt Ltd, Surat, Gujarat
  - Chopda Medicare & Research Centre Pvt. Ltd: Magnum Heart Institute, Nashik, Maharashtra
- Kenya (4):
  - KEMRI/CRDR, Siaya, KEMRI Clinical Research Annex, Kisumu, Siaya County
  - Gertrude's Children's Hospital, Nairobi
  - Kenya Medical Research Institute - Centre for Respiratory Disease Research, Nairobi
  - Center for Research In Therapeutic Sciences (CREATES), Strathmore University Medical Centre, Nairobi
- Nigeria (3):
  - University College Hospital Ibadan, Ibadan, Oyo/ibadan North
  - Aminu Kano Teaching Hospital, Kano
  - Lagos University Teaching Hospital, Lagos
- United Kingdom (2):
  - University Hospitals Bristol and Weston NHS Foundation Trust, Bristol
  - Bristol Royal Infirmary, Bristol

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Li Z, Alt C, Dufu K, Hutchaleelaha A, Xu Q, Zhang X, Li CM, Rademacher P, Bosmajian C, Pochron MP, Partridge JR, Oksenberg D, Cathers BE. Discovery of Osivelotor (GBT021601): A Potent, Next-Generation Sickle Hemoglobin Polymerization Inhibitor. ACS Med Chem Lett. 2025 Jul 8;16(8):1526-1532. doi: 10.1021/acsmedchemlett.5c00076. eCollection 2025 Aug 14. PMID 40832524
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=GBT021601-021